CLINICAL TRIAL: NCT02650687
Title: Optimizing Postoperative Cognition the Elderly
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 13-1692; 1K23AG048332-01A1 (NIH)
Record Dates: First submitted 2015-12-23; First posted 2016-01-08 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Cognitive Dysfunction; POCD
Keywords: Postoperative Cognitive Dysfunction; Elderly, geriatric; Anesthesia; Anesthetic depth; Bispectral index monitor; Function; Recovery after surgery; Surgery
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Brain Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elective Non Cardiac Surgical Patients: 65 years of age and older
  Interventions: Procedure: Processed EEG

INTERVENTIONS:
Procedure: Processed EEG — In the operating room. Processed EEG will be measured using the Bispectral Index (BIS) monitor which is standard of care.
  Other Names: brain waves

SUMMARY:
This study will recruit surgical patients more than 65 years old. Patients who participate will wear a sticker on their forehead during surgery which monitors their brain waves (electroencephalogram, EEG) and participate in memory testing before and after surgery. Brain wave patterns will be compared between patients who have problems with memory and thinking after surgery and those who do not. The hypothesis is that there will be characteristic brain wave patients for who will go on to have problems with memory and thinking after surgery.

DETAILED DESCRIPTION:
Eligible patients will be identified through the computerized scheduling system at the Icahn School of Medicine at Mount Sinai. After informed consent, patients will complete cognitive and tests at least one but not more than 30 days prior to surgery. In the recovery room the Post Anesthesia Recovery Scale (PQRS), and CAM-ICU delirium screening will be administered. Immediate recovery will be recorded using the Postoperative Recovery Scale (PQRS) on postoperative day 1 and 3, and 1 week.

Longterm functional recovery will be measured with the Alzheimer's Disease Research Center (ADRC) Instrumental Activities for Daily Living (IADL-24). Postsurgical complications will be recorded including unplanned ICU admissions, postoperative myocardial infarction and stroke (risk less than 1 % in most cases), wound infection and reoperation. The full cognitive and functional battery will be repeated at 3 months and 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older
* having major elective non-cardiac surgery requiring general anesthesia requiring at least a 2 day hospital stay

Exclusion Criteria:

* previous diagnosis of dementia, stroke, cardiac or intracranial surgery
* inability to consent or communicate in English or Spanish
* major uncorrected hearing or vision deficit, Parkinson's disease, or major psychiatric disease which will be determined by phone interview and computer medical records abstracted by the primary investigator.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Eligible patients will be identified through the computerized scheduling system at the Icahn School of Medicine at Mount Sinai.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2015-10; Primary Completion 2019-02-25 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
UDS battery | 3 months
  Postoperative Cognitive Dysfunction - UDS battery is the standard ADRC neuropsychological battery and will be used to measure cognition

SECONDARY OUTCOMES:
Processed EEG | 1 year
  Processed EEG will be measured using the Bispectral Index (BIS) monitor.
CAM-ICU | baseline
  The Confusion Assessment Method-ICU is a delirium screening tool for Intensive Care Unit (ICU) patients, assessing 4 features: alteration/fluctuation in mental status, Inattention, altered level of consciousness, and disorganized thinking.
CAM-ICU | Day 1
  The Confusion Assessment Method-ICU is a delirium screening tool for Intensive Care Unit (ICU) patients, assessing 4 features: alteration/fluctuation in mental status, Inattention, altered level of consciousness, and disorganized thinking.
CAM-ICU | Day 3
  The Confusion Assessment Method-ICU is a delirium screening tool for Intensive Care Unit (ICU) patients, assessing 4 features: alteration/fluctuation in mental status, Inattention, altered level of consciousness, and disorganized thinking.
CAM-ICU | 1 week
  The Confusion Assessment Method-ICU is a delirium screening tool for Intensive Care Unit (ICU) patients, assessing 4 features: alteration/fluctuation in mental status, Inattention, altered level of consciousness, and disorganized thinking.
PQRS | baseline
  Short -Term Recovery: Postoperative Quality of Recovery Scale (PQRS)
PQRS | Day 1
  Short -Term Recovery: Postoperative Quality of Recovery Scale (PQRS)
PQRS | Day 3
  Short -Term Recovery: Postoperative Quality of Recovery Scale (PQRS)
PQRS | 1 week
  Short -Term Recovery: Postoperative Quality of Recovery Scale (PQRS)
UDS battery | 1 year
  Postoperative Cognitive Dysfunction - UDS battery is the standard ADRC neuropsychological battery and will be used to measure cognition

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Deiner, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Dustin Boone M, Lin HM, Liu X, Kim J, Sano M, Baxter MG, Sieber FE, Deiner SG. Processed intraoperative burst suppression and postoperative cognitive dysfunction in a cohort of older noncardiac surgery patients. J Clin Monit Comput. 2022 Oct;36(5):1433-1440. doi: 10.1007/s10877-021-00783-0. Epub 2021 Dec 3. PMID 34862586
- [Derived] Cooter Wright M, Bunning T, Eleswarpu SS, Heflin MT, McDonald SR, Lagoo-Deenadalayan S, Whitson HE, Martinez-Camblor P, Deiner SG, Berger M. A Processed Electroencephalogram-Based Brain Anesthetic Resistance Index Is Associated With Postoperative Delirium in Older Adults: A Dual Center Study. Anesth Analg. 2022 Jan 1;134(1):149-158. doi: 10.1213/ANE.0000000000005660. PMID 34252066
- [Derived] Esses GJ, Liu X, Lin HM, Khelemsky Y, Deiner S. Preoperative frailty and its association with postsurgical pain in an older patient cohort. Reg Anesth Pain Med. 2019 May 6:rapm-2018-100247. doi: 10.1136/rapm-2018-100247. Online ahead of print. PMID 31061107
- [Derived] Deiner S, Liu X, Lin HM, Sieber F, Boockvar K, Sano M, Baxter MG. Subjective cognitive complaints in patients undergoing major non-cardiac surgery: a prospective single centre cohort trial. Br J Anaesth. 2019 Jun;122(6):742-750. doi: 10.1016/j.bja.2019.02.027. Epub 2019 Apr 17. PMID 31003631